CLINICAL TRIAL: NCT05840250
Title: Improving Glucose Control and Self-Management in Adults With Type 2 Diabetes From Health Disparate Groups Using Continuous Glucose Monitoring and Education Support
Brief Title: Continuous Glucose Monitoring and Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: shortage in the availability on the continuous glucose monitor making it unable to reopen enrollement
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2022-0402
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Diabetes
Keywords: Glucose Control; Type 2 Diabetes; Continuous Glucose Monitoring; Educational support
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Glucose Monitoring and Education Support Group (Experimental): Participants will be provided with a device to monitor their blood glucose (Abbott Free Style Libre2 Flash CGM system) along with educational materials to better understand and manage their diabetes and other supporting services. Pre and post intervention surveys will be implemented. Participants will be closely monitored for 3 months and then followed up for 3 more months for a total of 6-month participation.
  Interventions: Other: Continuous Glucose Monitoring and Education Support

INTERVENTIONS:
Other: Continuous Glucose Monitoring and Education Support — Participants will be provided with a device to monitor their blood glucose (Abbott Free Style Libre2 Flash CGM system) along with educational materials to better understand and manage their diabetes and other supporting services. Pre and post intervention surveys will be implemented. Participants will be closely monitored for 3 months and then followed up for 3 more months for a total of 6-month participation.

SUMMARY:
The study is a longitudinal single-arm prospective study design. Adult patients who are African American or Hispanic with type 2 diabetes mellitus will be recruited to participate in this study. The goal of the study is to determine if the use of a continuous glucose monitoring system will improve diabetes management in persons from health disparity background.

The subjects will be closely monitored for the first 3 months as they utilize the continuous glucose monitor and engage in diabetes education classes. They will then be followed for an additional 3 months to determine if they are able to maintain the same glucose control as experienced for the initial 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with type 2 diabetes mellitus ≥18 years
* African-American or Hispanic
* with A1c ≥8% to ≤12%

Exclusion Criteria:

* Patients with type 1 diabetes,
* pregnant,
* End-Stage Renal Disease,
* recent use of any CGM within the last 12 months,
* on steroid therapy and history of adhesive allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
A1c - Marker of overall glucose control | At 3 months post enrollment
  A1c levels measured at 12 weeks post enrollment will be compared to the baseline A1c level (measured at enrollment).
A1c - Marker of overall glucose control | At 6 months post enrollment
  A1c levels measured at 24 weeks post enrollment will be compared to the baseline A1c level (measured at enrollment).
Glycemic control | At 3 months post enrollment
  To investigate the effect of the Continuous Glucose Monitoring (CGM) device and educational support on the Glycemic control. Glycemic control will be measured based on the percent time that glucose is on target vs off target. On target is within the normal range of 70-180 mg/dL. Off target includes: <54 mg/dL (critical low glucose); < 70 mg/dL (low glucose); >180 mg/dL (high glucose); and >250 mg/dL (very high).
  The range at 12 weeks post enrollment will be compared to the baseline data that will be collected after the first 14 days (2 weeks).
Glycemic control | At 6 months post enrollment
  To investigate the effect of the Continuous Glucose Monitoring (CGM) device and educational support on the Glycemic control. Glycemic control will be measured based on the percent time that glucose is on target vs off target. On target is within the normal range of 70-180 mg/dL. Off target includes: <54 mg/dL (critical low glucose); < 70 mg/dL (low glucose); >180 mg/dL (high glucose); and >250 mg/dL (very high).
  The range at 24 weeks post enrollment will be compared to the baseline data that will be collected after the first 14 days (2 weeks).

SECONDARY OUTCOMES:
Blood pressure | At 3 months post enrollment
  To determine if CGM and diabetes education affects Blood pressure. Blood pressure will be measured before the CGM/education begins and at the 3 month follow up appointment.
Weight | At 3 months post enrollment
  To determine if CGM and diabetes education affects weight. Weight will be measured before the CGM/education begins and at the 3 month follow up appointment.
BMI | At 3 months post enrollment
  To determine if CGM and diabetes education affects BMI. BMI will be calculated before the CGM/education begins and at the 3 month follow up appointment.
ER visit | For the 3 months post enrollment
  To determine if CGM and diabetes education glycemic control as demonstrated by ER visit due to hypoglycemia or hyperglycemic events.
Hospital admissions | For the 3 months post enrollment
  To determine if CGM and diabetes education glycemic control as demonstrated by hospital admission due to hypoglycemia or hyperglycemic events.
Glycemic control - Episodes of hypoglycemia | For the 3 months post enrollment
  To determine if CGM and diabetes education glycemic control as demonstrated by the number of episodes of hypoglycemia occurred during the 3 months post enrollment.
  The number of hypoglycemic events will be recorded at baseline (2 weeks) and compared to the data collected at the 12 weeks timepoint.
Diabetes knowledge | At 3 months post enrollment
  To determine if CGM and diabetes education Diabetes knowledge. Diabetes knowledge will be measured before the CGM/education begins (baseline) and at the 3 month follow up appointment. Diabetes knowledge will be measured using a 10-item survey called "The SKILLD Knowledge Assessment Scale" (Spoken Knowledge in Low Literacy patients with Diabetes (SKILLD)). The scale ranges from 0% to 100% with higher scores demonstrating better knowledge.
Diabetes self-care | At 3 months post enrollment
  To determine if CGM and diabetes education affects Diabetes self-care. Diabetes self-care will be measured before the CGM/education begins (baseline) and at the 3 month follow up appointment. Diabetes self-care will be measured using a 11-item survey and reflects on activities for the past 7 days. The survey used is called "Summary of Diabetes Self-Care Activities" . The survey includes five regimen areas: Diet, Exercise, Blood-Glucose Testing, Foot-Care, and Smoking Status and each area is scored separately based on the number of days an event took place (from 0 for 0 days to 7 for each day).
Diabetes distress | At 3 months post enrollment
  To determine if CGM and diabetes education affects Diabetes distress. Diabetes distress will be measured before the CGM/education begins (baseline) and at the 3 month follow up appointment. Diabetes distress will be measured using a survey. The 17-item survey called "Diabetes Distress Screening (DDS17)" assesses the difficulties living with diabetes as it relates to disease.
  management, support, emotional burden and access to care. Each item is scored from 1 (No distress) to 6 (distress). The overall score is calculated as the mean of all items and higher the number the higher the distress level reported.
Satisfaction with CGM device | At 3 months post enrollment
  Using a satisfaction scale, the satisfaction with the CGM device will be measured at 3 months post enrollment. A 15-item Survey will be used to evaluate treatment burden/satisfaction with using a continuous glucose monitor. The survey contains four subscales (Openness, Emotional Burden, Behavioral Burden, and Worthwhileness) as well as a total score. Each can be obtained by calculating the mean item response score for the groups of items below. Each item is scored between 1 and 5 with 1 being strongly disagree and 5 being strongly agree. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Colette Knight, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golden SH, Brown A, Cauley JA, Chin MH, Gary-Webb TL, Kim C, Sosa JA, Sumner AE, Anton B. Health disparities in endocrine disorders: biological, clinical, and nonclinical factors--an Endocrine Society scientific statement. J Clin Endocrinol Metab. 2012 Sep;97(9):E1579-639. doi: 10.1210/jc.2012-2043. Epub 2012 Jun 22. PMID 22730516
- [Background] Hill-Briggs F, Adler NE, Berkowitz SA, Chin MH, Gary-Webb TL, Navas-Acien A, Thornton PL, Haire-Joshu D. Social Determinants of Health and Diabetes: A Scientific Review. Diabetes Care. 2020 Nov 2;44(1):258-79. doi: 10.2337/dci20-0053. Online ahead of print. No abstract available. PMID 33139407
- [Background] Bergenstal RM, Kerr MSD, Roberts GJ, Souto D, Nabutovsky Y, Hirsch IB. Flash CGM Is Associated With Reduced Diabetes Events and Hospitalizations in Insulin-Treated Type 2 Diabetes. J Endocr Soc. 2021 Feb 2;5(4):bvab013. doi: 10.1210/jendso/bvab013. eCollection 2021 Apr 1. PMID 33644623
- [Background] Haak T, Hanaire H, Ajjan R, Hermanns N, Riveline JP, Rayman G. Flash Glucose-Sensing Technology as a Replacement for Blood Glucose Monitoring for the Management of Insulin-Treated Type 2 Diabetes: a Multicenter, Open-Label Randomized Controlled Trial. Diabetes Ther. 2017 Feb;8(1):55-73. doi: 10.1007/s13300-016-0223-6. Epub 2016 Dec 20. PMID 28000140
- [Background] Vigersky RA, Fonda SJ, Chellappa M, Walker MS, Ehrhardt NM. Short- and long-term effects of real-time continuous glucose monitoring in patients with type 2 diabetes. Diabetes Care. 2012 Jan;35(1):32-8. doi: 10.2337/dc11-1438. Epub 2011 Nov 18. PMID 22100963
- [Background] Rodriguez JE, Campbell KM. Racial and Ethnic Disparities in Prevalence and Care of Patients With Type 2 Diabetes. Clin Diabetes. 2017 Jan;35(1):66-70. doi: 10.2337/cd15-0048. No abstract available. PMID 28144049
- [Background] Yaron M, Roitman E, Aharon-Hananel G, Landau Z, Ganz T, Yanuv I, Rozenberg A, Karp M, Ish-Shalom M, Singer J, Wainstein J, Raz I. Effect of Flash Glucose Monitoring Technology on Glycemic Control and Treatment Satisfaction in Patients With Type 2 Diabetes. Diabetes Care. 2019 Jul;42(7):1178-1184. doi: 10.2337/dc18-0166. Epub 2019 Apr 29. PMID 31036546
- [Background] Martens T, Beck RW, Bailey R, Ruedy KJ, Calhoun P, Peters AL, Pop-Busui R, Philis-Tsimikas A, Bao S, Umpierrez G, Davis G, Kruger D, Bhargava A, Young L, McGill JB, Aleppo G, Nguyen QT, Orozco I, Biggs W, Lucas KJ, Polonsky WH, Buse JB, Price D, Bergenstal RM; MOBILE Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Patients With Type 2 Diabetes Treated With Basal Insulin: A Randomized Clinical Trial. JAMA. 2021 Jun 8;325(22):2262-2272. doi: 10.1001/jama.2021.7444. PMID 34077499
- [Background] Karter AJ, Parker MM, Moffet HH, Gilliam LK, Dlott R. Association of Real-time Continuous Glucose Monitoring With Glycemic Control and Acute Metabolic Events Among Patients With Insulin-Treated Diabetes. JAMA. 2021 Jun 8;325(22):2273-2284. doi: 10.1001/jama.2021.6530. PMID 34077502
- [Background] Haak T, Hanaire H, Ajjan R, Hermanns N, Riveline JP, Rayman G. Use of Flash Glucose-Sensing Technology for 12 months as a Replacement for Blood Glucose Monitoring in Insulin-treated Type 2 Diabetes. Diabetes Ther. 2017 Jun;8(3):573-586. doi: 10.1007/s13300-017-0255-6. Epub 2017 Apr 11. PMID 28401454
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Polonsky WH, Fisher L, Hessler D, Edelman SV. Development of a New Measure for Assessing Glucose Monitoring Device-Related Treatment Satisfaction and Quality of Life. Diabetes Technol Ther. 2015 Sep;17(9):657-63. doi: 10.1089/dia.2014.0417. Epub 2015 Apr 29. PMID 25923812
- [Background] Rothman RL, Malone R, Bryant B, Wolfe C, Padgett P, DeWalt DA, Weinberger M, Pignone M. The Spoken Knowledge in Low Literacy in Diabetes scale: a diabetes knowledge scale for vulnerable patients. Diabetes Educ. 2005 Mar-Apr;31(2):215-24. doi: 10.1177/0145721705275002. PMID 15797850
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Gal RL, Cohen NJ, Kruger D, Beck RW, Bergenstal RM, Calhoun P, Cushman T, Haban A, Hood K, Johnson ML, McArthur T, Olson BA, Weinstock RS, Oser SM, Oser TK, Bugielski B, Strayer H, Aleppo G. Diabetes Telehealth Solutions: Improving Self-Management Through Remote Initiation of Continuous Glucose Monitoring. J Endocr Soc. 2020 Jun 23;4(9):bvaa076. doi: 10.1210/jendso/bvaa076. eCollection 2020 Sep 1. PMID 32864542
- [Background] Vigersky R, Shrivastav M. Role of continuous glucose monitoring for type 2 in diabetes management and research. J Diabetes Complications. 2017 Jan;31(1):280-287. doi: 10.1016/j.jdiacomp.2016.10.007. Epub 2016 Oct 14. PMID 27818105